CLINICAL TRIAL: NCT05304754
Title: Phase I / II Study on Infusion of Alloreactive or Stimulated Natural Killer Cells With IL-15 ex Vivo After Haploidentical Transplantation of Hematopoietic Progenitors in Pediatric Patients With Hematological Neoplasms
Brief Title: "Phase I / II Study on Infusion of Natural Killer Cells After Haploidentical Transplantation in Pediatric Patients"
Acronym: PHINK
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHINK -01/2019; 2019-000911-10 (EudraCT Number)
Record Dates: First submitted 2022-01-12; First posted 2022-03-31 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: High-risk Leukemias
MeSH Terms: interventions — Interleukin-15

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- KIR mismatch aloreactive NK donor cells (Active Comparator): Three patients from each cohort will receive NK aloreactive cells from a KIR mismatch donor
  Interventions: Biological: Alloreactive NK cells
- NK cells stimulated ex vivo with IL-15 from KIR match donor (Experimental): Three patients in each cohort will receive ex vivo stimulated NK cells with IL-15 from a KIR match donor.
  Interventions: Biological: NK cells stimulated ex vivo with IL-15

INTERVENTIONS:
Biological: NK cells stimulated ex vivo with IL-15 — When patient and donor are KIR-HLA match, the patient submits all HLA class I molecules, or in the absence of any, your donor does not have this molecule, or having it lacks the corresponding KIR receiver. For more information detailed information on the product under investigation, reference is made to the Dossier of the Research Product (IMPD): PEI 09-008
  Arms: NK cells stimulated ex vivo with IL-15 from KIR match donor
Biological: Alloreactive NK cells — When the patient lacks the HLA class I molecule and his donor has this molecule and also the donor NK cells have the KIR receptor that recognizes the absence of the corresponding HLA class I ligand
  Arms: KIR mismatch aloreactive NK donor cells

SUMMARY:
Phase I / II study on infusion of alloreactive or stimulated Natural Killer cells with IL-15 ex vivo after haploidentical transplantation of hematopoietic progenitors in pediatric patients with hematologic malignancies (PHINK

DETAILED DESCRIPTION:
Haploidentical hematopoietic stem cell transplantation (haploTPH) constitutes a highly complex but effective procedure for some hematologic malignancies high-risk pediatric patients in the absence of an identical HLA donor. Relapse Post-transplant leukemia is the main problem for survival. Just like reported different expert groups on haploTPH in adults and children, there is a determining role of Natural Killer (NK) cells in haploTPH as inducers powerful graft-versus-leukemia (EIcL) effect. The presence of NK cells allo-reactive is correlated with a lower relapse rate, in addition to favoring the graft, decrease graft versus recipient disease (GVHD) and decrease viral infections. This only occurs in half of the donor-recipient pairs, so that, in its absence, it is necessary to develop other strategies for activating the NK cells. In this sense, the investigational group has extensive experience in research translational with NK cells and is a pioneer in infusing ex vivo activated NK cells with IL-15.

The investigators propose a phase I / II clinical trial with dose escalation, multicenter, framed in the Spanish Group of Hematopoietic Transplantation / Marrow Transplant Bone in Children (GETH / GETMON), to determine the safety and efficacy of a post-haploTPH IL-15 alloreactive / stimulated NK cell infusion in children with malignant blood diseases. The investigators will monitor immune reconstitution, chimerism, Post-transplantation NK cell expansion, phenotype, and function.

Secondarily evaluate the effectiveness of therapy on the incidence of graft failure; EICR; viral reactivations; transplant-related mortality; and relapse of leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes with age ≤ 21 years.
* Not having an identical HLA donor (family or non-family) available in the time needed for the donation of hematopoietic parents.
* Having a haploidenic donor available
* Diagnosis of high-risk hematological malignancy. This includes:
* i. High risk ALL in first complete remission (RC1);
* ii. ALL in second complete remission (RC2);
* iii. ALL in third complete remission (RC3) or later;
* iv. High risk AML in RC1;
* v. AML in RC2 or later;
* vi. Relapsed AML with <25% blasts in bone marrow;
* vii. AML related to previous treatments in CR> 12 months;
* viii. Primary or secondary myelodysplastic syndrome
* ix. NK cell leukemia, biphenotypic or undifferentiated in RC1 or later,
* x. Chronic myeloid leukemia (CML) in accelerated phase, in chronic phase with persistent molecular positivity, or with intolerance to tyrosine kinase inhibitors
* xi. Hodgkin's lymphoma in RC2 or later after failure of autologous TPH, or unable to mobilize hematopoietic progenitors for autologous TPH
* xii. Non-Hodgkin's lymphoma in RC2 or later after failure of autologous TPH, or unable to mobilize hematopoietic progenitors for autologous TPH
* xiii. Myelomonocytic juvenile leukemia.
* Positive pre-transplant evaluation
* i. Left ventricular ejection fraction > 40% or shortening fraction ≥ 25%;
* ii. Creatinine clearance (ACr) or glomerular filtration rate (TFG) ≥ 50 ml/min/1.73 m2
* iii. Forced Vital Capacity (FVC) ≥ 50% of predicted value or pulse-oximetry ≥ 92% if the patient cannot perform the pulmonary function tests;
* iv. Karnofsky or Lansky Index (depending on the patient's age) ≥ 50;
* v. Bilirubin ≤ 3 times the upper limit of normal for age
* vi. Alanine aminotransferase (ALT) ≤ 5 times the upper limit of normal for age
* vii. Women who are not breastfeeding.
* viii. No uncontrolled bacterial, fungal, or viral infections at the time of inclusion.
* Women of childbearing potential must have a negative serum or urine pregnancy test performed within 14 days prior to trial inclusion and must agree to use highly effective contraceptive methods (diaphragms plus spermicide or male condom plus spermicide, oral contraceptive combined with a second method of contraceptive implant, injectable contraceptive, permanent intrauterine device, sexual abstinence, or partner with vasectomy) during study participation and for six months after the last trial visit. In the case of male patients with reproductive capacity, they must commit to using an appropriate barrier method for the duration of the study and for up to 6 months thereafter

Exclusion Criteria:

* Patients with an active infectious process or other serious underlying medical condition
* Patients who, according to the investigator's criteria, have a history of poor compliance with therapy.
* Patients who after a psycho-social evaluation are advised as not suitable for the procedure:
* i. Social-family situation that makes correct participation in the study impossible.
* ii. Patients with emotional or psychological problems secondary to the illness such as post-traumatic stress disorder, phobias, delusions, psychosis, with the need for support from specialists.
* iii. Evaluation of the involvement of family members in the health of the patient
* Inability to understand the information about the trial
* Received an investigational drug within 30 days prior to the start of therapy or within 5 half-lives of receiving an investigational drug, whichever is longer.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (TLD) | 52 weeks
  To determine dose-limiting toxicity (TLD) of a single infusion of aloreactive NK cells or ex vivo IL-15-stimulated NK cells after haploTPH in pediatric patients with high-risk leukemias.
Maximum tolerated dose (MTD) | 52 weeks
  To determine maximum tolerated dose (MTD) of a single infusion of aloreactive NK cells or ex vivo IL-15-stimulated NK cells after haploTPH in pediatric patients with high-risk leukemias.

SECONDARY OUTCOMES:
Efficacy of post haploTPH NK cell therapy | Week 52
  The efficacy of post haploTPH NK cell therapy will be determined, comparing it with the historical cohort recently reported by GETH/GETMON in the incidence of graft failure, acute/chronic GVHD, viral reactivations (CMV, EBV, HHV-6, adenovirus, BKV), transplant-related mortality (TRM), and leukemia relapse.
Clinical evolution of patients | Week 52
  The clinical course of patients will be compared based on the dose of infused NK cells, KIR match vs. KIR mismatch NK cells, expansion, chimerism, and phenotypic and functional characteristics of the infused NK cells, and the speed and characteristics of immune reconstitution post haploTPH.
Monitor immune reconstitution and characterize NK cells | Week 52
  Immune reconstitution will be monitored by quantifying immunoglobulins at different times, and characterizing NK cells in patients, at a phenotypic and functional level, for 1 year after haploTPH

CONTACTS AND LOCATIONS:
Locations (10):
- Spain (10):
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Infantil Universitario Niño Jeús, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Málaga (Carlos de Haya), Málaga
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario La Fe, Valencia

REFERENCES:
- [Background] Ciceri F, Labopin M, Aversa F, Rowe JM, Bunjes D, Lewalle P, Nagler A, Di Bartolomeo P, Lacerda JF, Lupo Stanghellini MT, Polge E, Frassoni F, Martelli MF, Rocha V; Acute Leukemia Working Party (ALWP) of European Blood and Marrow Transplant (EBMT) Group. A survey of fully haploidentical hematopoietic stem cell transplantation in adults with high-risk acute leukemia: a risk factor analysis of outcomes for patients in remission at transplantation. Blood. 2008 Nov 1;112(9):3574-81. doi: 10.1182/blood-2008-02-140095. Epub 2008 Jul 7. PMID 18606875
- [Background] Ruggeri L, Capanni M, Urbani E, Perruccio K, Shlomchik WD, Tosti A, Posati S, Rogaia D, Frassoni F, Aversa F, Martelli MF, Velardi A. Effectiveness of donor natural killer cell alloreactivity in mismatched hematopoietic transplants. Science. 2002 Mar 15;295(5562):2097-100. doi: 10.1126/science.1068440. PMID 11896281
- [Background] Leung W, Iyengar R, Triplett B, Turner V, Behm FG, Holladay MS, Houston J, Handgretinger R. Comparison of killer Ig-like receptor genotyping and phenotyping for selection of allogeneic blood stem cell donors. J Immunol. 2005 May 15;174(10):6540-5. doi: 10.4049/jimmunol.174.10.6540. PMID 15879158
- [Background] Aversa F. Haploidentical haematopoietic stem cell transplantation for acute leukaemia in adults: experience in Europe and the United States. Bone Marrow Transplant. 2008 Mar;41(5):473-81. doi: 10.1038/sj.bmt.1705966. Epub 2008 Jan 7. PMID 18176612
- [Background] Lang P, Handgretinger R. Haploidentical SCT in children: an update and future perspectives. Bone Marrow Transplant. 2008 Oct;42 Suppl 2:S54-9. doi: 10.1038/bmt.2008.285. PMID 18978746
- [Background] Leung W, Campana D, Yang J, Pei D, Coustan-Smith E, Gan K, Rubnitz JE, Sandlund JT, Ribeiro RC, Srinivasan A, Hartford C, Triplett BM, Dallas M, Pillai A, Handgretinger R, Laver JH, Pui CH. High success rate of hematopoietic cell transplantation regardless of donor source in children with very high-risk leukemia. Blood. 2011 Jul 14;118(2):223-30. doi: 10.1182/blood-2011-01-333070. Epub 2011 May 25. PMID 21613256
- [Background] Handgretinger R, Chen X, Pfeiffer M, Mueller I, Feuchtinger T, Hale GA, Lang P. Feasibility and outcome of reduced-intensity conditioning in haploidentical transplantation. Ann N Y Acad Sci. 2007 Jun;1106:279-89. doi: 10.1196/annals.1392.022. Epub 2007 Apr 18. PMID 17442774
- [Background] Moretta A, Pende D, Locatelli F, Moretta L. Activating and inhibitory killer immunoglobulin-like receptors (KIR) in haploidentical haemopoietic stem cell transplantation to cure high-risk leukaemias. Clin Exp Immunol. 2009 Sep;157(3):325-31. doi: 10.1111/j.1365-2249.2009.03983.x. PMID 19664139
- [Background] Ciurea SO, Mulanovich V, Jiang Y, Bassett R, Rondon G, McMannis J, de Lima M, Shpall EJ, Champlin RE. Lymphocyte recovery predicts outcomes in cord blood and T cell-depleted haploidentical stem cell transplantation. Biol Blood Marrow Transplant. 2011 Aug;17(8):1169-75. doi: 10.1016/j.bbmt.2010.11.020. Epub 2010 Nov 30. PMID 21126598
- [Background] Leen AM, Christin A, Myers GD, Liu H, Cruz CR, Hanley PJ, Kennedy-Nasser AA, Leung KS, Gee AP, Krance RA, Brenner MK, Heslop HE, Rooney CM, Bollard CM. Cytotoxic T lymphocyte therapy with donor T cells prevents and treats adenovirus and Epstein-Barr virus infections after haploidentical and matched unrelated stem cell transplantation. Blood. 2009 Nov 5;114(19):4283-92. doi: 10.1182/blood-2009-07-232454. Epub 2009 Aug 21. PMID 19700662
- [Background] Distler E, Bloetz A, Albrecht J, Asdufan S, Hohberger A, Frey M, Schnurer E, Thomas S, Theobald M, Hartwig UF, Herr W. Alloreactive and leukemia-reactive T cells are preferentially derived from naive precursors in healthy donors: implications for immunotherapy with memory T cells. Haematologica. 2011 Jul;96(7):1024-32. doi: 10.3324/haematol.2010.037481. Epub 2011 Apr 12. PMID 21486863
- [Background] Miller JS, Soignier Y, Panoskaltsis-Mortari A, McNearney SA, Yun GH, Fautsch SK, McKenna D, Le C, Defor TE, Burns LJ, Orchard PJ, Blazar BR, Wagner JE, Slungaard A, Weisdorf DJ, Okazaki IJ, McGlave PB. Successful adoptive transfer and in vivo expansion of human haploidentical NK cells in patients with cancer. Blood. 2005 Apr 15;105(8):3051-7. doi: 10.1182/blood-2004-07-2974. Epub 2005 Jan 4. PMID 15632206
- [Background] Triplett BM, Horwitz EM, Iyengar R, Turner V, Holladay MS, Gan K, Behm FG, Leung W. Effects of activating NK cell receptor expression and NK cell reconstitution on the outcomes of unrelated donor hematopoietic cell transplantation for hematologic malignancies. Leukemia. 2009 Jul;23(7):1278-87. doi: 10.1038/leu.2009.21. Epub 2009 Feb 12. PMID 19212329
- [Background] Ciurea SO, Schafer JR, Bassett R, Denman CJ, Cao K, Willis D, Rondon G, Chen J, Soebbing D, Kaur I, Gulbis A, Ahmed S, Rezvani K, Shpall EJ, Lee DA, Champlin RE. Phase 1 clinical trial using mbIL21 ex vivo-expanded donor-derived NK cells after haploidentical transplantation. Blood. 2017 Oct 19;130(16):1857-1868. doi: 10.1182/blood-2017-05-785659. Epub 2017 Aug 23. PMID 28835441
- [Background] Wanquet A, Bramanti S, Harbi S, Furst S, Legrand F, Faucher C, Granata A, Calmels B, Lemarie C, Picard C, Chabannon C, Weiller PJ, Castagna L, Blaise D, Devillier R. Killer Cell Immunoglobulin-Like Receptor-Ligand Mismatch in Donor versus Recipient Direction Provides Better Graft-versus-Tumor Effect in Patients with Hematologic Malignancies Undergoing Allogeneic T Cell-Replete Haploidentical Transplantation Followed by Post-Transplant Cyclophosphamide. Biol Blood Marrow Transplant. 2018 Mar;24(3):549-554. doi: 10.1016/j.bbmt.2017.11.042. Epub 2017 Dec 13. PMID 29247781
- [Background] Perez-Martinez A, Fernandez L, Valentin J, Martinez-Romera I, Corral MD, Ramirez M, Abad L, Santamaria S, Gonzalez-Vicent M, Sirvent S, Sevilla J, Vicario JL, de Prada I, Diaz MA. A phase I/II trial of interleukin-15--stimulated natural killer cell infusion after haplo-identical stem cell transplantation for pediatric refractory solid tumors. Cytotherapy. 2015 Nov;17(11):1594-603. doi: 10.1016/j.jcyt.2015.07.011. Epub 2015 Sep 1. PMID 26341478
- [Background] Perez-Martinez A, Iyengar R, Gan K, Chotsampancharoen T, Rooney B, Holladay M, Ramirez M, Leung W. Blood dendritic cells suppress NK cell function and increase the risk of leukemia relapse after hematopoietic cell transplantation. Biol Blood Marrow Transplant. 2011 May;17(5):598-607. doi: 10.1016/j.bbmt.2010.10.019. Epub 2010 Oct 25. PMID 20977942
- [Background] Van Elssen CHMJ, Ciurea SO. NK cell therapy after hematopoietic stem cell transplantation: can we improve anti-tumor effect? Int J Hematol. 2018 Feb;107(2):151-156. doi: 10.1007/s12185-017-2379-x. Epub 2017 Dec 1. PMID 29196968
- [Background] Vela M, Corral D, Carrasco P, Fernandez L, Valentin J, Gonzalez B, Escudero A, Balas A, de Paz R, Torres J, Leivas A, Martinez-Lopez J, Perez-Martinez A. Haploidentical IL-15/41BBL activated and expanded natural killer cell infusion therapy after salvage chemotherapy in children with relapsed and refractory leukemia. Cancer Lett. 2018 May 28;422:107-117. doi: 10.1016/j.canlet.2018.02.033. Epub 2018 Feb 23. PMID 29477379
- [Background] Fernandez L, Leivas A, Valentin J, Escudero A, Corral D, de Paz R, Vela M, Bueno D, Rodriguez R, Torres JM, Diaz-Almiron M, Lopez-Collazo E, Martinez-Lopez J, Perez-Martinez A. How do we manufacture clinical-grade interleukin-15-stimulated natural killer cell products for cancer treatment? Transfusion. 2018 Jun;58(6):1340-1347. doi: 10.1111/trf.14573. Epub 2018 Mar 14. PMID 29542132